CLINICAL TRIAL: NCT06383351
Title: Perception and Impact on Oral Health-related Quality of Life of Peri-implant Diseases. A Cross-sectional Study
Brief Title: Patients' Illness Perception of Peri-implant Diseases. A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Associate Professor, University of Siena
Other Study IDs: BQ001
Record Dates: First submitted 2024-04-16; First posted 2024-04-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Peri-implant Mucositis; Perception; Survey; Questionnaires; Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peri-implant disease patients: Patients with a diagnosis of peri-implant mucositis or peri-implantitis
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Two sets of questionnaires will be administered to patients:
  * Questionnaire about their perception of peri-implant disease (Brief Illness Perception Questionnaire; 9 questions, answers will be registered on a scale of 0 to 10);
  * Oral Health Impact Profile 14 (OHIP-14) questionnaire.

SUMMARY:
Despite extensive research on periodontitis, little attention has been given to the symptoms and perception of peri-implant diseases and their impact on oral health-related quality of life. The study aims to assess patient perception of these diseases and their impact on quality of life through a cross-sectional observational study. Patients will be recruited from the Unit of Periodontics at "Le Scotte" University Hospital and will undergo diagnosis followed by questionnaire assessments. No follow-up visits are planned, and validated questionnaires will be administered to evaluate perception and impact on quality of life. Study procedures will include recording biometric peri-implant parameters and administering questionnaires such as the Brief Illness Perception Questionnaire (BIPQ) and Oral Health Impact Profile-14 (OHIP-14).

DETAILED DESCRIPTION:
Peri-implant diseases are inflammatory processes, influenced by biofilm, affecting the soft and hard tissues surrounding dental implants. They encompass two main conditions: peri-implant mucositis and peri-implantitis. While professional biofilm removal, coupled with plaque control, is considered the gold standard treatment, its efficacy is limited. Therefore, enhancing prevention and early diagnosis strategies for peri-implant complications is crucial. Despite extensive research on patient perception of periodontitis symptoms, little attention has been given to the symptoms and perception of peri-implant diseases and their impact on oral health-related quality of life. This observational study aims to assess patient perception of peri-implant diseases and their impact on oral health-related quality of life (OHRQoL). The study is a cross-sectional observational study. Patients will be recruited from the Unit of Periodontics, Department of Medical Biotechnologies, at "Le Scotte" University Hospital. Following diagnosis of peri-implant disease, patients meeting inclusion and exclusion criteria specified in the protocol will be included. Given the study's cross-sectional nature, no follow-up visits are planned. Validated questionnaires regarding the perception and impact on the quality of life of peri-implant diseases will be administered. Study procedures will include recording biometric parameters extracted from a complete periodontal examination and administering questionnaires on the perception and impact on the quality of life of peri-implant diseases: Brief Illness Perception Questionnaire (BIPQ) and Oral Health Impact Profile-14 (OHIP-14).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old;
* Presence of at least one dental implant;
* Presence of bleeding and/or suppuration upon probing of the peri-implant mucosa;
* Ability and willingness to provide written consent for participation in the study.

Exclusion Criteria:

* Pregnancy or breastfeeding status;
* Patients unable to communicate in Italian or English;
* Inability to perform proper oral hygiene maneuvers;
* Inability or unwillingness to provide written consent for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited consecutively from those attending the Unit of Periodontics, Departoment of Medical Biotechnologies, at "Le Scotte" University Hospital (Siena, Italy).
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Assessment of patient's perception of their peri-implant disease through the Brief Illness Perception Questionnaire (Brief IPQ) | Baseline
  Brief Illness Perception Questionnaire consists of 9 questions, each one evaluated on a scale of 0 to 10 (minimum score of 0, maximum score of 90). Higher scores mean a higher patient's perception of the disease (higher scores mean worse outcome).
Assessment of peri-implant disease's impact on the oral health-related quality of life through the Oral Health Impact Profile 14. | Baseline
  14 questions about the impact of oral health on the quality of life; each question will be evaluated on a scale of 1 to 5 (minimum score of 0, maximum score of 70). Higher scores mean that patient's oral health impacts more significantly on their quality of life (higher scores, worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Discepoli, DDS, MsC, PhD, Principal Investigator — Department of Medical Biotechnologies, University of Siena
Locations (1):
- AOUS, Siena, Italy

REFERENCES:
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Machado V, Botelho J, Ramos C, Proenca L, Alves R, Cavacas MA, Mendes JJ. Psychometric properties of the Brief Illness Perception Questionnaire (Brief-IPQ) in periodontal diseases. J Clin Periodontol. 2019 Dec;46(12):1183-1191. doi: 10.1111/jcpe.13186. Epub 2019 Oct 21. PMID 31446628
- [Background] Discepoli N, Marruganti C, Mirra R, Pettinari G, Ferrari Cagidiaco E, Ferrari M. Patients' illness perception before and after non-surgical periodontal therapy: A pre-post quasi-experimental study. J Periodontol. 2022 Jan;93(1):123-134. doi: 10.1002/JPER.21-0052. Epub 2021 May 25. PMID 33997985
- [Derived] De Rubertis I, Fratini A, Ferrari A, Mirra R, Discepoli N. Cognitive and Emotional Peri-Implant Diseases Perception in a Cohort of Periodontitis Patients: A University-Based Cross-Sectional Study. J Clin Periodontol. 2025 Nov;52(11):1573-1583. doi: 10.1111/jcpe.70011. Epub 2025 Aug 18. PMID 40827002